CLINICAL TRIAL: NCT05630534
Title: Study of Minocycline Accelerated Intracerebral Hemorrhage Absorption (MACHA)
Brief Title: Minocycline Accelerates Intracerebral Hemorrhage Absorption
Acronym: MACHA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); The Second Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHZhejiangULiMin
Record Dates: First submitted 2022-11-06; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Intracerebral Hemorrhage
Keywords: Minocycline; hematoma absorption
MeSH Terms: conditions — Cerebral Hemorrhage; cyclopia sequence | interventions — Minocycline; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): This intervention arm will receive oral or intranasal minocycline capsules 100 mg Q12H, first dose 200 mg, start on the fifth day of cerebral hemorrhage, for 14 days
  Interventions: Drug: Minocycline
- Control（starch） (Placebo Comparator): This arm will receive oral or intranasal administration of identically packaged placebo capsules (starch) 100 mg Q12H, first dose 200 mg, start on the fifth day of cerebral hemorrhage, for 14 days
  Interventions: Other: starch

INTERVENTIONS:
Drug: Minocycline — Minocycline is a tetracycline antibiotic routinely used in clinical practice for the treatment of bacterial infection and acne.
  Other Names: Minomycin
  Arms: Minocycline
Other: starch — Use starch capsules as placebo
  Arms: Control（starch）

SUMMARY:
Minocycline has been found to reduce cerebral edema secondary to cerebral hemorrhage, promote hematoma absorption, and shorten hematoma absorption time; clinical studies have been conducted to confirm the safety in the treatment, but no significant hematoma absorption effect was seen with short duration of drug use. Therefore, the investigators propose to conduct a multicenter randomized controlled clinical trial to determine its accelerating effect on hematoma absorption.

DETAILED DESCRIPTION:
There is a significant increase in the incidence of spontaneous intracerebral hemorrhage, combined with a high mortality rate. Surgical treatment is mainly used to remove intracerebral hematoma with a supratentorial volume greater than 20ml, and most intracerebral hematomas below 20mL are left to absorb on their own, and the absorption time of such hematomas is about 4 to 6 weeks. Minocycline is a tetracycline antibiotic routinely used in clinical practice for the treatment of bacterial infection and acne.

It has been found that it can not only reduce iron overload after intracerebral hemorrhage and inhibit neuroinflammation, but also reduce secondary cerebral edema. Some animal experiments have confirmed that it can promote hematoma absorption through iron chelation and shorten hematoma absorption time; clinical studies have been conducted to confirm the safety in the treatment of intracerebral hemorrhage, but no significant effect has been seen with short duration of drug use. No clinical RCT study has been conducted to confirm its accelerating effect on the absorption of adult intracerebral hematoma. Therefore, the investigators propose to conduct a multicenter randomized controlled clinical trial to determine its accelerating effect on hematoma absorption, and this study will have important clinical practical value.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Spontaneous intracerebral hemorrhage by CT scan
* Intracerebral hematoma volume is less than 16ml
* No surgical treatment of hematoma evacuation

Exclusion Criteria:

* Allergies to tetracycline antibiotics
* Pregnancy or suspected pregnancy (pregnancy test will be done on women with fertility potential)
* Hepatic and/or renal insufficiency
* Glasgow Coma Scale of 5 or less
* Secondary cerebral hemorrhage caused by trauma, arteriovenous malformation, aneurysm, tumor or other reasons
* Thrombocytopenia (platelet count<75000/mm3) or coagulation dysfunction (INR>1.4)
* Incapable to take care of themselves in past life (score of Rankin scale before stroke>2)
* Signed DNR (Do Not Resuscitate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in modified Rankin Scale score at 90 days of onset | 90 days
  modified Rankin Scale score (points ranging from 0 to 6)

SECONDARY OUTCOMES:
Number adverse events related to minocycline within 90 days | 90 days
  nausea, vomiting, C-diff, hepatic toxicity, dermatitis, anaphylaxis, renal injury, fever

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No
Keep the IPD, if other researchers need the data, they can email the investigator.